CLINICAL TRIAL: NCT04884750
Title: Community-based Design and Evaluation of A Conversational Agent to Promote SARS-COV2 Vaccination in Black Churches
Brief Title: Conversational Agent Vaccine Promotion RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northeastern University (Other)
Collaborators: Boston University (Other); Boston Medical Center (Other); Georgia Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB#18-07-02
Record Dates: First submitted 2021-05-05; First posted 2021-05-13 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Pandemics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High engagement mechanisms, tailed content (Experimental): During this time the investigators will conduct a 2x2 factorial RCT (with the individual the unit of random assignment and measurement) to assess the impact of two app design features on engagement and outcomes: (1) the investigators will manipulate engagement mechanisms (ENGAGEMENT), including reminder notifications and trust-building dialogue by the ECA and, (2) independently manipulate cultural tailoring of vaccination promotion counseling language used by the agent (TAILORING) to either adaptive religiosity (tailored) or secular (non-tailored). The investigators' primary hypotheses are that participants with have significantly greater vaccination completion rates in the high engagement and tailored conditions at 6 months (H1) and 12 months (H2) compared to other conditions.
  Interventions: Behavioral: ECA-ACE Vaccination Promotion Intervention
- Low engagement mechanisms, tailed content (Experimental): manipulate low engagement mechanisms while provide adaptive religiosity (tailored) content
  Interventions: Behavioral: ECA-ACE Vaccination Promotion Intervention
- High engagement mechanism, non-tailed content (Experimental): manipulate high engagement mechanisms while provide secular (non-tailored) content
  Interventions: Behavioral: ECA-ACE Vaccination Promotion Intervention
- Low engagement mechanism, non-tailed content (Experimental): manipulate low engagement mechanisms and provide secular (non-tailored) content
  Interventions: Behavioral: ECA-ACE Vaccination Promotion Intervention

INTERVENTIONS:
Behavioral: ECA-ACE Vaccination Promotion Intervention — A smartphone-based embodied conversational agent that educates users and motivates them to obtain vaccinations for SARS-CoV-2 and Influenza, according to Boston Public Health Commission guidelines.

SUMMARY:
The objective of this study is to assess the use of and satisfaction with the ECA intervention over a 12-month period, its ability to increase SARS-CoV-2 and influenza vaccination in the BMATP community, and the comparative effectiveness of proactive engagement strategies and cultural tailoring on these factors. The Investigators will assess app use and satisfaction among these participants, along with self-reported vaccination attitudes and behavior, at 6 months and 12 months.

During this time the investigators will conduct a 2x2 factorial RCT (with the individual the unit of random assignment and measurement) to assess the impact of two app design features on engagement and outcomes: (1) the investigators will manipulate engagement mechanisms (ENGAGEMENT), including reminder notifications and trust-building dialogue by the ECA and, (2) independently manipulate cultural tailoring of vaccination promotion counseling language used by the agent (TAILORING) to either adaptive religiosity (tailored) or secular (non-tailored). The investigators' primary hypotheses are that participants with have significantly greater vaccination completion rates in the high engagement and tailored conditions at 6 months (H1) and 12 months (H2) compared to other conditions. The investigators' secondary hypotheses are that participants will use the app more, be more satisfied with the ECA, be more advanced in their stage of change, and have greater knowledge, self-efficacy, and decisional-balance from baseline to 6 and 12 months, in the high engagement and tailored conditions. In addition to the RCT participants, all members of the 12 participating BMATP churches will be invited to use the app (via snowball recruitment), to increase the utility of the social networking functions of the app by having as many users as possible.

DETAILED DESCRIPTION:
4.1.a.1. Randomization. Study participants will be randomized into one of the four study conditions (ENGAGEMENT x TAILORING) using blocked randomization with randomly permuted block sizes of 2 and 4, by software on the central server referenced when participants first activate the app on their phone.

Participants will continue using the app at home, and will be called at 6 months and 12 months to assess outcome measures during a videoconference call with a research assistant.

4.1.a.2. Qualitative Interviews. The investigators will conduct interviews with a sample of participants completing the study (12), as well as with Church and Health Ministry leadership (12) to understand overall acceptance of ECA-ACE and barriers to deployment and use.

4.1.a.3. Qualitative Methods for all Project Focus Groups and Interviews. Videoconference-based focus groups and interviews will be facilitated using a semi-structured interview guide, audio-recorded, and transcribed verbatim by a professional transcription service. The investigators will conduct a thematic analysis of these transcripts guided by the investigators' research questions with the aim of identifying design insights. The investigators will use grounded theory analysis, including constant comparisons, axial and selective coding, and memo writing. Using NVivo 12.5.0 software, two researchers will inductively code transcripts separately, labeling emergent phenomena in the data to arrive at a codebook. Two researchers will then independently apply the codebook to participant transcripts, meeting regularly to discuss discrepancies in the applications of the codes, updates to the codebook, and contradictory data. Sample sizes specified should be adequate to reach thematic saturation relative to the investigators' research questions.

ELIGIBILITY:
Inclusion Criteria:

1. over 18 years old;
2. speaks English fluently;
3. is able to independently consent;
4. has adequate corrected vision to use the ECA system (based on a 1 minute ECA functional screener deployed over the web);
5. has adequate hearing to use the ECA system;
6. owns a recent model iPhone or Android smartphone.
7. do not meet current Boston Public Health commission guidelines for SARS-CoV-2 vaccination OR do not meet current Boston Public Health commission guidelines for Influenza vaccination.

Exclusion Criteria:

1. they are not able demonstrate comprehension of the research study;
2. they are unable to use the screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of SARS-CoV-2 vaccination status | baseline, 6months, 12months
  Vaccination completion will be assessed via self-report by asking whether participants are up-to-date with Boston Public Health Commission vaccination guidelines (yes or no) for SARS-CoV-2
Change of Influenza vaccination status Influenza vaccination status | baseline, 6months, 12months
  Vaccination completion will be assessed via self-report by asking whether participants are up-to-date with Boston Public Health Commission vaccination guidelines (yes or no) for Influenza

SECONDARY OUTCOMES:
Change of Satisfaction Status | 6 months, 12 months
  Self report System Usability Scale (self report), plus system use from log file analysis.
Stage of Change for Vaccination | baseline,6months,12months
  Self report of Precontemplation, Contemplation, Preparation, or Action/Maintenance for vaccination
Self-Efficacy for Vaccination | baseline,6months,12months
  Self report of confidence in ability to get vaccinated in light of barriers
Decisional Balance for Vaccination | baseline,6months,12months
  Self report of Pros and Cons of vaccination
Knowledge | baseline,6months,12months
  Knowledge of COVID-19 and Influenza assessed via 10-item true/false knowledge tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The dissemination plan has two overall goals:
  1. Scientific Dissemination of Study Findings
     For our scientific stakeholders, the investigators will publish findings in the peer-reviewed scientific literature, and also present findings at scientific conferences and through invited seminars to share these findings. In addition, the investigators plan to make data available for collaborative analyses with colleagues around the world.
  2. Community Dissemination of Intervention
  In the final two years of the effort, intervention materials will be revised based on feedback and lessons learned from the RCTs. The smartphone app will be opened so that anyone can download and use it, and extended to automatically collect basic sociodemographics, primary outcome measures, and usage directly from users if they electronically consent upon initiation of the app and saved to the central database, so that dissemination, use, and outcomes can be tracked and evaluated during dissemination.